CLINICAL TRIAL: NCT07286045
Title: Visual Assessment and Rapid On-Site Evaluation for Touch Imprints From Biopsy Tissue in Diagnosing Pleural Effusion Using Medical Thoracoscopy
Brief Title: Visual Assessment vs ROSE in Diagnosing Pleural Effusion Using Medical Thoracoscopy
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Fathi Elbagalaty MD, Lecturer of pulmonary medicine, Ain Shams University
Other Study IDs: FMASU R190/2024
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Thoracoscopy; Pleural Effusion Disorder
Keywords: pleural effusion , thoracoscopy
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pleural biopsy tissue blocks, histopathology slides, and touch-imprint cytology preparations collected during medical thoracoscopy. No genetic or genomic testing is planned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thoracoscopy patients: Participants are adults undergoing medical thoracoscopy for evaluation of undiagnosed pleural effusion or suspected pleural disease. All participants receive standard-of-care thoracoscopy with pleural biopsies. During the procedure, the thoracoscopist provides a visual assessment of the pleura, and touch-imprint cytology samples are obtained for Rapid On-Site Evaluation (ROSE). Final histopathology is used as the diagnostic reference standard.
  Interventions: Procedure: Medical thoracoscopy

INTERVENTIONS:
Procedure: Medical thoracoscopy — All participants undergo medical thoracoscopy, during which pleural surfaces are directly inspected, and targeted pleural biopsies are obtained as part of routine clinical care. During the procedure, the thoracoscopist records a gross visual impression of whether pleural findings appear benign or malignant. Touch-imprint cytology slides are prepared from biopsy samples and evaluated immediately using Rapid On-Site Evaluation (ROSE). Final histopathology of biopsy specimens serves as the diagnostic reference standard. No experimental treatments are given.

SUMMARY:
The goal of this observational diagnostic study is to find how well two evaluation methods used during medical thoracoscopy can help identify whether pleural disease is malignant or benign. The study focuses on adults undergoing thoracoscopy for undiagnosed pleural effusion or suspected pleural disease.

The main questions this study aims to answer are:

How accurate is the thoracoscopist's visual assessment of the pleura in predicting malignancy?

How accurate is Rapid On-Site Evaluation (ROSE) of touch-imprint cytology compared with final laboratory histopathology?

Researchers will compare thoracoscopic visual impressions with ROSE results to determine which method provides more reliable real-time diagnostic information.

Participants will:

Undergo medical thoracoscopy as part of their clinical evaluation.

Have pleural biopsy samples assessed on-site using ROSE.

Have standard histopathology testing performed for final diagnosis.

This study may help improve decision-making during thoracoscopy by identifying whether combining visual assessment with ROSE leads to faster and more accurate diagnosis of pleural disease.

DETAILED DESCRIPTION:
Pleural effusion is a common clinical problem, and distinguishing malignant from benign causes is crucial for guiding treatment. Medical thoracoscopy allows direct visualization of the pleural surfaces and enables targeted biopsies. Although experienced clinicians often rely on the gross appearance of pleural abnormalities, visual assessment alone can be limited by overlap between malignant and benign features. Rapid On-Site Evaluation (ROSE) of touch-imprint cytology has emerged as a technique that may provide immediate microscopic information during the procedure, potentially improving diagnostic accuracy and reducing the need for repeat procedures.

This observational study prospectively evaluated the diagnostic performance of thoracoscopic visual inspection compared with ROSE during medical thoracoscopy. Thirty-three adult patients undergoing thoracoscopy for undiagnosed pleural effusion or suspected pleural disease were included. During the procedure, the thoracoscopist recorded a visual impression of whether pleural findings appeared malignant or benign. Touch-imprint slides were prepared from pleural biopsy specimens and assessed immediately by a trained cytopathologist using ROSE. All biopsy samples were subsequently analyzed by formal histopathology, which served as the reference standard.

The study measured sensitivity, specificity, accuracy, predictive values, receiver operating characteristic (ROC) curves, and agreement using Cohen's kappa. Visual assessment showed high sensitivity but limited specificity. ROSE demonstrated high overall accuracy and strong agreement with final histopathology, suggesting it may substantially improve real-time diagnostic confidence. By integrating both visual inspection and ROSE, clinicians may achieve more reliable intraoperative decision-making and potentially streamline patient management during thoracoscopy.

ELIGIBILITY:
Inclusion criteria included adult patients (>18 years) with undiagnosed pleural effusion undergoing medical thoracoscopy.

Exclusion Criteria:

Exclusion Criteria, while Medical thoracoscopy is generally safe; patients with the following conditions were excluded in accordance with reported contraindications (Jin et al., 2020):

1. Absolute contraindications:

   * Refusal to participate in the study.
   * Extensive pleural adhesions (e.g., pleural fibrosis, post-infection, or prior pleurodesis).
   * Inadequate pleural space for thoracoscopy.
2. Relative contraindications**

   * Coagulopathy (platelet count <60 × 10⁹/L or INR >1.2), unless corrected prior to the procedure. The use of aspirin and clopidogrel was not considered a contraindication.
   * Inability to tolerate the lateral decubitus position.
   * Unstable hemodynamic status.
   * Severe hypoxemia requiring high-flow oxygen therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>18 years) with undiagnosed exudative pleural effusion undergoing medical thoracoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Rapid On-Site Evaluation (ROSE) and Visual assessment | Time Frame: During thoracoscopy (immediate assessment) with confirmation by final histopathology within 2-7 days
  ROSE: Touch-imprint cytology slides prepared from pleural biopsy specimens are evaluated on-site by a trained cytopathologist to classify pleural disease as malignant or benign.
  Thoracoscopic Visual Assessment: The thoracoscopist records a gross visual impression of the pleura as malignant or benign during the procedure.
  Outcome Metrics: Sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), overall accuracy, and area under the receiver operating characteristic curve (AUC) for each method compared with the reference standard of histopathology.
  Additional Analysis: Agreement between ROSE and histopathology will be quantified using Cohen's κ statistic.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Rationale: This study involves diagnostic observations collected during routine clinical care. Data contain potentially identifiable patient information and are intended for internal research use only

REFERENCES:
- [Background] Jin F, Wang H, Li Q, Li S, Lai G, Huang J, Huang Y, Jiang T, Bai C, Li S, Li W, Lu Y, Song Y, Sun R, Chen C, Zhang J, Zhang X, Zhou R, Zhou X, Chen Y, Du Y, Hu C, Zhou H. Expert consensus for diagnosis and treatment using medical thoracoscopy in China. J Thorac Dis. 2020 May;12(5):1799-1810. doi: 10.21037/jtd-19-2276. PMID 32642085
- [Background] Ahmed MI, El Hefny RA, Farhat ES. New challenge in double-bore medical thoracoscopy in Fayoum University Hospital. Egypt J Chest Dis Tuberc. 2024;73(1):37-43.